CLINICAL TRIAL: NCT05564923
Title: CARG, VES13, G8 Scales in Predicting Drug Toxicity in Patients Receiving Nivolumab
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Namik Kemal University (Other)
Responsible Party: Principal Investigator, Asoc. Prof. Erdoğan Selçuk Şeber, Asoc Prof., Namik Kemal University
Other Study IDs: NIVOTOXTOOL
Record Dates: First submitted 2022-09-02; First posted 2022-10-04 (Actual); Last update posted 2022-10-04 (Actual); Status verified 2022-10

CONDITIONS: Nivolumab Related Toxicity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- group 1: Advanced cancer patients over 65 years of age receiving nivolumab
  Interventions: Drug: there is no intervention

INTERVENTIONS:
Drug: there is no intervention — there is no intervention

SUMMARY:
The Geriatric 8 (G8), Vulnerable Elders Survey (VES-13), and Cancer and Aging Research Group (CARG) questionnaires are among the main tests whose purpose is to predict the risk of chemotherapy-induced toxicity (CRT) and allow treatment. Investigators aimed to investigate the effect of using the G8, VES13, and CARG scales in the geriatric age group in cancer patients receiving nivolumab treatment in predicting side effects.

DETAILED DESCRIPTION:
Investigator aimed to examine whether the G8, VES13, and CARG scales can shed light on clinicians in predicting side effects during the use of nivolumab in geriatric cancer patients. In the chemotherapy unit, demographic information, diagnosis date of the disease, previous treatments, comorbidities, and CARG, VES13, and G8 questionnaires will be recorded face-to-face to the patients who meet the study criteria. In addition, routine hemogram and biochemistry tests, which were requested by the patient's follow-up physician before Nivolumab treatment and which will be requested by the patient's own physician during follow-up visits, will be recorded prospectively. Side effects that may occur during nivolumab treatment will be pursued at each visit. CTCA v.6. will be used for grading.

inclusion criteria

1-Advanced cancer patients whose nivolumab treatment was started by the physician followed up (independent of diagnosis) 2-60 years and over, 3-ECOG performance score 0-1 4-Patients who signed the informed consent form

exclusion criteria

1. Under 60 years old
2. Ecog score >1

ELIGIBILITY:
Inclusion Criteria:

* Advanced stage cancer patients who have been treated with nivolumab
* be over 60 years old

Exclusion Criteria:

* be under the age of 60

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Advanced stage cancer patients who have been treated with nivolumab
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-09-02 (Actual); Primary Completion 2023-06-17 (Estimated); Study Completion 2023-08-17 (Estimated)

PRIMARY OUTCOMES:
grade 3-4 nivolumab toxicity | one year from first patient enrolled
  grading will be made according to the CTCA V.6

CONTACTS AND LOCATIONS:
Locations (1):
- Tekirdağ Namık Kemal University, Tekirdağ, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No